CLINICAL TRIAL: NCT07136428
Title: A Single Arm, Open-label Phase Ib/II Study of Asciminib in HER2+ Breast Cancer Brain Metastases (ASCENdANT)
Brief Title: Asciminib in HER2+ Breast Cancer Brain Metastases
Acronym: ASCENdANT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00117131
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HER2+ Metastatic Breast Cancer
MeSH Terms: interventions — asciminib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asciminib Trastuzumab (Experimental): Combination of asciminib and trastuzumab
  Interventions: Combination Product: Asciminib and Trastuzumab

INTERVENTIONS:
Combination Product: Asciminib and Trastuzumab — Each study treatment cycle will last 21 days. Asciminib will be taken orally every day during the treatment period at the dose determined as the MTD during the safety lead-in in combination with trastuzumab at a standard dose of 6mg/kg IV. Asciminib dose will begin at 80 mg daily (dose level 1), with a potential range from 40 mg daily (dose level -1A, with trastuzumab) to 200 mg bid (dose level 3, with trastuzumab) depending on the results of the safety lead-in. Trastuzumab will be given intravenously (IV) or subcutaneously (SQ) on Day 1 of each 21 day cycle.

SUMMARY:
The purpose of this study is to evaluate the intracranial response rate of a combination of asciminib/trastuzumab for the treatment of patients with metastatic HER2+ breast cancer with brain metastases.

DETAILED DESCRIPTION:
Despite recent advances in the HER2+ space, BrM remain incurable, are associated with significant morbidity, and remain an unmet medical need. Once patients develop resistance to the early-line HER2-directed agents, there are few effective therapies, especially for patients with BrM. ABL kinases are being considered as a potential strategy for treating metastatic cancers, including metastatic HER2+ BC and BrM. The drug asciminib (ABL001, Novartis), an allosteric ABL kinase inhibitor currently FDA approved for treatment of CML. In this single-arm, open label multi-center Phase Ib/II study, patients with stage IV HER2+ BCBrM with at least one progressive or new brain metastasis measuring >5mm will receive asciminib along with standard of care trastuzumab, first as part of a safety lead-in followed by a Phase 2 trial in 13 patients. A 4-15patient safety run-in will be initially conducted to determine the MTD of asciminib/trastuzumab combination therapy, or the maximal safe dose at which patients in the second part of the study will receive. There will be 4 dose levels of combination therapy in the safety run-in. DLTs will be monitored and dose mods will be executed as needed. The treatment period for this study will last for at least 9 cycles. Each cycle will last 21 days. Asciminib will be taken orally at the assigned dose every day during the treatment period. Trastuzumab will be given intravenously (IV) or subcutaneously (SQ) at the assigned dose on Day 1 of each 21 day cycle. Participants will continue on study therapy until disease progression, toxicity, or patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of consent
* Patients with HER2+ metastatic breast cancer with at least one progressive or new brain metastasis measuring >5mm; prior local therapy to other intracranial lesions allowed
* At least 1 prior standard of care therapy for metastatic disease
* Must have previously received T-DXd and Tucatinib. If a patient has not received T-DXd or Tucatinib as part of standard early line therapy due to allergies or intolerability, the requirement of prior T-DXd and Tucatinib treatment is waived.
* Participants must have adequate treatment washout period when applicable before enrollment, defined as:

  * >4 weeks from any major surgery
  * >1 week from any cranial radiation treatment
  * For cytotoxic containing agents, 5 half-lives or at least 21 days (whichever is shorter)
  * For weekly chemotherapy regimens, >2 weeks from chemotherapy; for every 3 weekly regimens, >3 weeks from chemotherapy. At least 2 weeks from other systemic or targeted or investigational therapies (other than endocrine therapy) for breast cancer. No washout is required for endocrine therapy (e.g. aromatase inhibitors, tamoxifen, fulvestrant) but patients should discontinue prior to start of protocol therapy.
  * Patients on ovarian suppression are allowed (but not required) to continue ovarian suppression at the discretion of their treating provider.
* Adequate organ function and bone marrow reserve as determined by the investigator
* Adequate hepatic and renal function and hematologic parameters:

  * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 9 g/dL
  * Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases are present)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated using the Cockcroft-Gault (CG) equation
* Left ventricular ejection fraction (LVEF) ≥ 50%.
* Females of childbearing potential must have a negative pregnancy test (serum or urine) at screening. If a pregnancy test using either method is positive or cannot be confirmed as negative, a second testing using the other method will be required for confirmation.
* Females of childbearing potential and males must be willing to abstain from heterosexual intercourse or to use highly effective contraception
* Can enroll with intracranial disease only; extracranial disease can be absent or non-measurable
* Focal leptomeningeal disease allowed at investigator discretion
* Performance status by Eastern Cooperative Oncology Group (ECOG) 0-2 (appendix 1)
* Written informed consent and HIPAA authorization for release of personal health information prior to enrollment. NOTE: HIPAA authorization may be included in the informed consent or obtained separately

Exclusion Criteria:

* No evidence of hemorrhage or impending herniation or need for immediate local therapy to intracranial disease or escalating dosing of steroids
* No grade 2 or greater peripheral neuropathy
* Diffuse and symptomatic leptomeningeal carcinomatosis
* Prolonged Qtc (QTcF>450), CHF or uncontrolled HTN
* Clinically significant cardiopulmonary disease.
* Acute or chronic pancreatitis within 6 months prior to first day of study treatment
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

  * tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice),
  * hepatitis B (known positive HBV surface antigen (HBsAg) result) ,
  * hepatitis C (note: hepatitis C testing at screening will only be performed on those at high risk or with known history), or
  * human immunodeficiency virus (positive HIV 1/2 antibodies) (note: HIV testing at screening will only be performed on those at high risk or with known history)
  * NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for ≥ 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.
* Unable for any reason to undergo MRI of the brain.
* Use of a strong cytochrome P450 (CYP)3A4 inhibitor within 5 half-lives of study treatment. .. Unable to avoid certain CYP3A4 or CYP2C9 substrates which cannot be co-administered with study treatment given altered substrate concentrations.
* Central nervous system exclusion - Based on screening brain MRI, patients must not have any of the following:

  * Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent)
  * Diffuse leptomeningeal disease or positive CSF cytology; however, discreet dural-based metastases are allowed
  * Poorly controlled seizures. Defined as seizures that continue to occur despite optimal anticonvulsant medications based on investigator discretion.
* Active infection requiring intravenous systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Patients with a prior or concurrent malignancy within last 5 years whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.
* Treatment with any investigational drug within 30 days prior to enrollment (Day 1 of study drug).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a dose-limiting toxicity at each dose level | Day 1 of treatment until 30 days post last dose
  Safety of administering asciminib in combination with trastuzumab by measuring number of participants with a dose-limiting toxicity at each dose level
Number of participants with a complete response (CR) or partial response (PR) | Day 1 of treatment through up to 112 weeks
  Efficacy at maximum tolerated dose (MTD) determined by the number of participants with a complete response (CR) or partial response (PR) as determined by Response Assessment in Neuro-Oncology (RANO) Criteria for Brain Metastases (RANO-BM).

SECONDARY OUTCOMES:
Median time to progression | Day 1 of treatment through up to 112 weeks
  Time to Progression (TTP) (both intracranial or extracranial) as determined by Response Assessment in Neuro-Oncology (RANO) Criteria for Brain Metastases (RANO-BM).
Progression Free Survival (PFS) | Day 1 of treatment through up to 110 weeks
  Progression free survival as determined by Response Assessment in Neuro-Oncology (RANO) Criteria for Brain Metastases (RANO-BM).
Overall Survival (OS) | Day 1 of treatment through up to 110 weeks
  Patients will be followed till death or off study due to any other reason.

IPD SHARING:
Plan to Share IPD: No